CLINICAL TRIAL: NCT01680302
Title: Effect of 3 Years of Exercise on Development of Atrial Fibrillation - A "Generation 100" Substudy
Brief Title: Effect of 3 Years of Exercise on Development of Atrial Fibrillation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/978b-2
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Prevention; Exercise
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High intensity exercise (Experimental): High intensity exercise(Borg 16) in intervals.
  Interventions: Behavioral: High intensity exercise
- Moderate intensity exercise (Experimental): Moderate intensity exercise 3 times a week.
  Interventions: Behavioral: Moderate intensity exercise
- Control group (Experimental): Exercise on their own. Follow current guidelines.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: High intensity exercise
  Arms: High intensity exercise
Behavioral: Moderate intensity exercise
  Arms: Moderate intensity exercise
Behavioral: Control — Advised to follow current guidelines for physical activity, but exercise on their own.
  Arms: Control group

SUMMARY:
This is a substudy of "Generation 100". In that study, 4000 healthy persons between 70 and 75 will be randomised to a moderate intensity training group, a high intensity training group or control group, with 3 years of exercise. The investigators will follow these persons and register all who develop atrial fibrillation during these 3 years, and at follow-up after ended intervention to see if there is differences in the number of persons who develop atrial fibrillation in the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the "Generation 100" study

Exclusion Criteria:

-

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1567 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of persons who develop atrial fibrillation during the 3 year intervention period | 3 years
  People who already have the diagnosis before randomisation will not be counted.

SECONDARY OUTCOMES:
Number of persons who develop atrial fibrillation during the 6 years after randomisation | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paal Loennechen, PhD, Study Chair — St. Olavs Hospital
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway